CLINICAL TRIAL: NCT03417986
Title: An Open-label, Multicenter, Controlled Pharmaco-dynamic Clinical Trial to Explore the the Amyloid Beta Draining Effect of Thiethylperazine (TEP) in Subjects With Newly Diagnosed Early-to-mild Dementia Due to Alzheimer's Disease in Comparison to Healthy Volunteers
Brief Title: Clinical Trial to Explore the the Amyloid Beta Draining Effect of Thiethylperazine (TEP) in Subjects With Newly Diagnosed Early-to-mild Dementia Due to Alzheimer's Disease (AD) in Comparison to Healthy Volunteers
Acronym: drainAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Immungenetics AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMU-AD-001
Record Dates: First submitted 2017-11-29; First posted 2018-01-31 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Alzheimer Disease
Keywords: Thiethylperazine; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — tetraethylpyrazine; Thiethylperazine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1a: TEP 26 mg daily for 4d (Experimental)
  Interventions: Drug: TEP
- Group 1b: TEP 52 mg daily for 4d (Experimental)
  Interventions: Drug: TEP
- Group 2: TEP 26 mg daily for 54d (Experimental)
  Interventions: Drug: TEP

INTERVENTIONS:
Drug: TEP — For safety reasons the clinical trial will first enroll 14 subjects (7 patients and 7 healthy volunteers) for Group 1a receiving 26 mg TEP daily for 4 days with subsequent safety evaluation, based on adverse events and the safety parameters discussed in the protocol. A second set of patients (Group 1b), which will receive a higher dosage of 52 mg per day for 4 days will be enrolled optionally after recommendation to continue and subsequently treatment Group 2 with a treatment paradigm of 26 mg TEP daily for 54 days will start.
  Subjects eligible for participation are subjects with newly diagnosed (within last 12 month) early-to-mild dementia due to AD and healthy volunteers who fulfill all inclusion criteria and have none of the exclusion criteria present at screening.
  Other Names: Thiethylperazine

SUMMARY:
This proof-of-mechanism clinical trial study will test the efficacy and safety of thiethylperazine (TEP) in subjects with early onset of Alzheimer's Disease (AD). There is a strong scientific rationale for this study: TEP is a very well-known substance that has been available since 1961 and approved for the prevention and treatment of nausea, vomiting as well as vertigo. Therefore, it has a well understood pharmacologic background and promising safety data. Using AD mouse models, it has been recently discovered and confirmed that TEP promotes transport of toxic Aβ from the brain into the blood. More importantly, it has also been demonstrated to improve learning deficits in mice. The striking biological effect of TEP in preclinical testing and its known safety and toxicity profile encourages the investigators to investigate this in a multicenter clinical trial in subjects with early-to-mild AD in comparison to healthy volunteers. The investigators will assess whether TEP is able to enhance the transport of Aβ peptides from the brain into the blood in subjects with early-to-mild AD and improves cognitive efficacy.

ELIGIBILITY:
Inclusion Criteria:

For AD subject

1. Newly diagnosed (< 12 months) early-to-mild Alzheimer's disease as classified by a Mini-Mental State Examination (MMSE) Score of 25-18 reconfirmed at screening
2. AD diagnosis confirmed by recommended examinations in accordance with German DGN (Deutsche Gesellschaft für Neurologie)/DGPPN (Deutsche Gesellschaft für Psychiatrie und Psychotherapie,Psychosomatik und Nervenheilkunde) S3 Guideline "Dementia" and to standard at the clinical unit by:

   * psychometric and cognitive tests
   * lumbar puncture in subjects with uncertain AD diagnosis following central nervous system (CNS) imaging
   * Clinical Dementia Rating (global CDR) is 0.5 or 1. Memory box score must be at least 0.5. Isolated or predominant episodic memory deficit, manifested as memory performance in the Logical Memory subscale (Delayed Paragraph Recall) from the Wechsler Memory Scale-III 1 below age adjusted norms, according to hospital standard)
3. AD subject has full legal competence according to investigator opinion
4. Ability to comply with requirements or cognitive and other testing for the entire length of the trial available

   For healthy volunteer
5. Subject is a non-demented volunteer, based on the assessment of medical history, physical examination and clinically laboratory data at screening as determined by the Investigator

   For AD subject and healthy volunteer
6. Age > 55 - < 75 years
7. Written informed consent to participate within this trial
8. Subject is on stable dose for at least 3 month prior to screening when receiving protocol-allowed concomitant medications at screening (e.g. acetylcholinesterase inhibitors, NMDA (N-methyl-D-aspartate) receptor antagonists)
9. For subject receiving anticholinergic agents, oral corticosteroids, propranolol, clonidine, antihistamines other than cetirizin and EBSTEL® a washout period of 4 weeks prior to screening must be completed. Concerning anticholinergic agents in Group 1a: only for high- to medium-potency anticholinergic agents a washout period of 4 weeks prior to screening must be completed.
10. Post-menopausal females (post menopausal amenorrhea for at least 2 years or surgically sterilized (hysterectomy), tubal ligation is not acceptable)
11. Male subjects with reproductive potential, and have not been surgically sterilized, that have been informed and agreed to that he and his partner must use a highly effective method of contraception (Pearl Index <1%) such as implants, injectables, combined oral contraceptives, or hormonal intrauterine devices (IUDs), or refrain from sexual intercourse during the trial and until 3 months after completion of the trial
12. Good general health with no additional disease states that could interfere with the trial due to the investigator's assessment

Exclusion Criteria:

Exclusion Criteria to be checked at Screening Visit:

1. CSF cut-off values identified during routine Neurochemical Dementia Diagnostics
2. History or evidence of other significant neurological disease of the Central Nervous System (such as Parkinson's disease, multi-infarct dementia, fronto-temporal dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supra nuclear palsy, epilepsy, myasthenia gravis, subdural hematoma or multiple sclerosis)
3. History of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities
4. Significant neuroimaging abnormalities, previously known or discovered on the MRI scan, including evidence of infection, infarction (> 3 mm in size), brain tumors (other than small meningiomas), or other focal lesions, multiple lacunas or lacunas in a critical memory structure or severe confluent microvascular disease (but not mild white matter changes, which are frequent with aging)
5. History or evidence of moderate congestive heart failure defined by the New York Heart Association criteria (class I-IV)
6. Clinical relevant ECG findings, abnormalities, e.g. pro-arrhythmic potential/effects on QT interval (QTc >450 msec for males, >470 msec for females, confirmed by manual assessment of ECG parameters)
7. History of new cardiovascular event within the last 6 months
8. Resting sitting vital signs: Systolic blood pressure ≤ 100 mmHg or ≥ 165 mmHg, Diastolic blood pressure ≤ 60 mmHg or ≥ 100 mmHg, heart rate ≤ 50 beats/min or ≥ 90 beats/min9. Clinically significant renal disease or insufficiency, including but not limited to creatinine value of >1.5 mg/dl
9. Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), total bilirubin, or alkaline phosphatase >2.5 times the upper limit of normal laboratory range, or history of severe hepatobiliary disease (e.g. hepatitis B or C, or cirrhosis) without enzyme elevation
10. Positive tested for hepatitis B surface antigen (HBsAG) or hepatitis C virus/antibodies (anti-HCV) for the first time within the last 6 months prior to the Screening Visit
11. Positive tested for human immunodeficiency virus (HIV) at Screening Visit
12. Fasting triglycerides >2.5 times of the upper limit of normal
13. Uncontrolled diabetes (FBG > 150 mg/dl)
14. Coagulopathy or any kind of anti-coagulant therapy
15. Extrapyramidal syndrome
16. Elevation of prolactin, e.g. subject with prolactin-dependent breast cancer or pituitary tumor
17. History of severe psychiatric disease like psychotic disorder or current anxiolytic or neuroleptic therapy (for dementia-related or other psychiatric disorder) within the last 3 months of enrolment
18. Chronic depression or bipolar disorder or history of major depression within the past 2 years or history of any episode of treatment-resistant depression (requiring > 1 antidepressants, Electroconvulsive Therapy (ECT) etc.)
19. Significant history of alcohol abuse or drug abuse within the past 6 months (at the judgment of the investigator)
20. Current treatment with TEP or treatment up to 24 month prior to screening
21. Known incompatibility of TEP or phenothiazines
22. Subject is receiving the following treatment that may interact with TEP, e.g. adrenaline, tricyclic antidepressants, narcotics, bromocriptine, MAO (monoamine oxidase) inhibitors, CYP2D6 inhibitors, tramadol, pentetrazol, levodopa, anticonvulsants, medication causing extrapyramidal symptoms increases the likelihood of central nervous system side effects
23. Participation in a clinical trial involving another investigational drug within 4 weeks prior to screening visit
24. Women of child bearing potential or women who are pregnant or nursing
25. Male subjects with reproductive potential who refuse to use adequate means of contraception during and up to 3 months after stopping treatment with TEP

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Efflux of Amyloid beta peptides (Group mean changes from baseline) | Gr. 1a: up to 10 days; Gr.1b / 2: up tp 84 days
  To demonstrate a significantly increased efflux of Amyloid beta peptides from the brain into the bloodstream in subjects with newly diagnosed (within last 12 month) early-to-mild dementia due to Alzheimer's Disease vs. healthy volunteers that is expected to be caused by the ABCC1 transporter-stimulating effect of thiethylperazine.

SECONDARY OUTCOMES:
Scores obtained in psychometric tests [Cognition] | Group 1a and 1b and Group 2 on day 1, day 10 (Groups 1a/b) day 14 (Group 2) and day 84 (End of Trial-Group 1b/2).
  Changes in scores obtained in psychometric tests in newly diagnosed (within last 12 month) subjects with early-to-mild dementia due to AD vs. healthy volunteers as well as the analysis of their changes from baseline will be determined after treatment with thiethylperazine.
Incidence of Treatment-Emergent Adverse Events [Safety and tolerability] | Gr. 1a: up to 10 days; Gr.1b / 2: up tp 84 days
  To assess the safety and tolerability of thiethylperazine in newly diagnosed (within last 12 month) subjects with early-to-mild dementia due to AD and to compare this profile with the outcome of a control group of healthy volunteers
  Assessments:
  Treatment-emergent Adverse Events (AEs) Treatment-emergent Serious Adverse Events (SAEs) Adverse Events leading to premature discontinuation of trial medication
Cerebrospinal fluid (CSF) levels of Tau | Gr. 1a: up to 10 days; Gr.1b / 2: up tp 84 days
  To investigate the effect of thiethylperazine on CSF levels of phosphoTau181 and total Tau in subjects with newly diagnosed (within last 12 month) early-to-mild dementia due to AD

CONTACTS AND LOCATIONS:
Overall Officials: Lutz Frölich, Prof. Dr., Principal Investigator — Zentralinstitut für seelische Gesundheit, Medizinische Fakultät Mannheim, Universität Heidelberg,
Locations (2):
- Germany (2):
  - Klinik für Psychiatrie und Psychotherapie Universitätsmedizin Göttingen, Göttingen
  - Zentralinstitut für seelische Gesundheit, Medizinische Fakultät Mannheim, Universität Heidelberg,, Mannheim